CLINICAL TRIAL: NCT07215533
Title: Differential Effects of HIIT vs. TRE on Type 2 Diabetes Risk in Youth and Younger Adults
Brief Title: Effects of HIIT vs. TRE on Type 2 Diabetes Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-435
Record Dates: First submitted 2025-04-28; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Obesity and Type 2 Diabetes; Metabolic Diseases; High-intensity Interval Training; Time-restricted Eating
Keywords: High-intensity Interval Training; Time-restricted Eating; Obesity; Type 2 Diabetes; Youth; Young Adults
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Metabolic Diseases; Intermittent Fasting | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity interval training (Experimental): HIIT: The 4-week HIIT intervention will use a stationary bicycle performed 3 times/week (a total of 12 sessions over the 4-week), performing at the CRL. All participants will perform a 20-minute HIIT protocol (20 repetitions of 10-seconds work time followed by 50-seconds resting/active recovery for the first two weeks, and 10 repetitions of 20-seconds work time followed by 100-seonds resting/active recovery for the rest of two weeks; targeted 90% HRmax) after 5-minute warm-up (10% HRmax). The supervisor (PI: Joon Young Kim and/or Graduate researcher: Wonhee Cho) will provide encouragement and supervision for exercise adherence. Heart rate (Polar, Polar Electro Oy, Kempele, Finland) and rating of perceived exertion (RPE; detail described in the questionnaire section) will be recorded.
  Interventions: Behavioral: High-intensity interval training
- Time-restricted eating (Experimental): Participants randomized into the TRE group will be instructed to consume all their calories within a 10-hour period. We will instruct participants that they can choose their time-window (early TRE [7am - 5pm] or late TRE [1pm - 11pm]), but it must remain constant for the duration of the study. Further, we will give no restrictions on the type of foods and/or the quantities individuals can consume. We will ask individuals to maintain their diet for the duration of the study. Participants will be given clear instructions on their diet and how to use the "MyFitnessPal" application. Participants will have their total daily energy requirement calculated using the following formula (Basal metabolic rate [BMR] x activity level) and will be told to eat that amount within their allotted time window. BMR will be calculated when participants have their body composition taken by the InBody. Participants will be told to start their 4-week diet the following day after visit.
  Interventions: Behavioral: Time-restricted eating
- Control Group (No Intervention): Participants randomized into the control group will be told to maintain their daily lifestyle and dietary habits for the duration of the four weeks.

INTERVENTIONS:
Behavioral: High-intensity interval training — The 4-week HIIT intervention will use a stationary bicycle performed 3 times/week (a total of 12 sessions over the 4-week), performing at the CRL. All participants will perform a 20-minute HIIT protocol (20 repetitions of 10-seconds work time followed by 50-seconds resting/active recovery for the first two weeks, and 10 repetitions of 20-seconds work time followed by 100-seonds resting/active recovery for the rest of two weeks; targeted 90% HRmax) after 5-minute warm-up (10% HRmax). The supervisor (PI: Joon Young Kim and/or Graduate researcher: Wonhee Cho) will provide encouragement and supervision for exercise adherence. Heart rate (Polar, Polar Electro Oy, Kempele, Finland) and rating of perceived exertion (RPE; detail described in the questionnaire section) will be recorded.
  Other Names: HIIT
  Arms: High-intensity interval training
Behavioral: Time-restricted eating — Participants randomized into the TRE group will be instructed to consume all their calories within a 10-hour period. We will instruct participants that they can choose their time-window (early TRE [7am - 5pm] or late TRE [1pm - 11pm]), but it must remain constant for the duration of the study. Further, we will give no restrictions on the type of foods and/or the quantities individuals can consume. We will ask individuals to maintain their diet for the duration of the study. Participants will be given clear instructions on their diet and how to use the "MyFitnessPal" application. Participants will have their total daily energy requirement calculated using the following formula (Basal metabolic rate [BMR] x activity level) and will be told to eat that amount within their allotted time window. BMR will be calculated when participants have their body composition taken by the InBody. Participants will be told to start their 4-week diet the following day after visit.
  Arms: Time-restricted eating

SUMMARY:
The primary aim of this randomized controlled trial is to examine the effects of a 4-week high-intensity interval training (HIIT) and time-restricted eating (TRE) intervention on cardiometabolic biomarkers in adolescents and young adults.

DETAILED DESCRIPTION:
As of 2015, an estimated 2 billion individuals were overweight (body mass index [BMI] ≥ 25 kg/m2), and one-third of them were obese (BMI ≥ 30 kg/m2). Obesity has become a serious health concern due to its related comorbidities, including cardiovascular disease (CVD) and type 2 diabetes (T2D). While adolescents and young adults are considered low risk for the development of CVD, individuals with obesity are still at a greater risk of CVD development than individuals without obesity. Changes to dietary and fitness habits are currently the first-line recommendations for preventing weight gain and improving cardiometabolic health in adolescents and young adults.

Caloric restriction (CR), which involves reducing caloric intake by up to 50% of normal daily calorie intake, is a common dietary intervention approach for weight management and improving cardiometabolic health in adolescents and adults with obesity.9 However, studies have shown that CR is hard to maintain, and individuals tend to regain the weight after the intervention is completed. Time-restricted eating (TRE) has been proposed as an alternative to calorie restriction (CR). TRE, a type of short-term fasting, is defined as periods of no caloric intake followed by periods of ad libitum (as much as desired) caloric intake. The fact that TRE does not intentionally limit energy intake, whereas CR does, could make it more appealing to individuals in terms of adherence, acceptability, and efficacy. TRE is an effective strategy in reducing body fat percentage and waist circumference in adolescents and adults with obesity.

Moreover, high-intensity interval training (HIIT), which involves repeating short periods of intense activity followed by low-intensity breaks, has been shown to be effective in improving cardiometabolic health (including lipids, blood pressure, and insulin sensitivity) in adults with obesity compared to other traditional exercises. In addition to its benefits on cardiometabolic health, previous studies have suggested that HIIT can be a time-efficient strategy to enhance body composition and cardiopulmonary fitness in adults with obesity.1

However, it is unknown if TRE or HIIT will produce a greater improvement in cardiometabolic health. Therefore, the goal of this study is to examine the independent effect of a 4-week TRE and HIIT intervention on cardiometabolic biomarkers in youth and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (age 14-17 years old with sex- and race-specific BMI percentile ≥85th) and young adults with overweight and obesity (age 18 to 30 years old with BMI ≥25 kg/m2)

Exclusion Criteria:

* Chronic medical conditions: heart disease, arrhythmias, diabetes, thyroid disease, bleeding disorder, history of pulmonary disease, hypertension, hepatorenal disease, musculoskeletal disorder, neuromuscular/neurological disease, autoimmune disease, cancer, peptic ulcers, anemia, or chronic infection (HIV).
* Have taken any heart, pulmonary, thyroid, anti-hyperlipidemic, hypoglycemic, anti- hypertensive, endocrinologic (e.g., thyroid, insulin, etc.), emotional/psychotropic (e.g., Prednisone, Ritalin, Adderall), neuromuscular/neurological, or androgenic medications (anabolic steroids).
* Have a pacemaker.

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Weight (kg) | Baseline and after 4 weeks of intervention
  Weight is measured in kilograms (kg) using a calibrated digital scale.
Height (cm) | Baseline and after 4 weeks of intervention
  Height is measured in centimeters (cm) using a wall-mounted stadiometer.
Body Mass Index (BMI) | Baseline and after 4 weeks of intervention
  Weight and height will be combined to report BMI in kg/m².
Waist Circumference and Hip Circumference | Baseline and after 4 weeks of intervention
  Waist and hip circumferences are measured while participants stand straight with their arms extended outward. A non-elastic tape measure is wrapped around the waist and hip, and measurements are taken to the nearest centimeter (cm).
Blood Lipid Profile | Baseline and after 4 weeks of intervention
  Blood lipid profile, including total cholesterol (TC), triglycerides (TG), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C), and fasting glucose (FG) are measured in milligrams per deciliter (mg/dL) using the Cholestech LDX Analyzer. Blood samples are obtained via fingerstick, with the first drop wiped away and the second drop collected for analysis. Participants stand or sit comfortably during collection. After blood collection, the site is cleaned and covered with gauze and a bandage as needed. This procedure is minimally invasive and typically causes little discomfort.
Blood Pressure | Baseline and after 4 weeks of intervention
  Systolic blood pressure (SBP) and diastolic blood pressure (DBP) are measured in millimeters of mercury (mmHg), and resting heart rate (RHR) is measured in beats per minute (bpm) using an automated blood pressure monitor. Participants sit quietly for five minutes with minimal movement prior to measurement. A cuff is placed on the right upper arm (bicep area), and the monitor initiates inflation, deflation, and reinflation cycles. Participants are instructed not to move during the measurement process. All equipment is disinfected before and after each use with antiviral, antibacterial, and antifungal disposable wipes by a researcher wearing gloves.
Carotid-Femoral Pulse Wave Velocity | Baseline and after 4 weeks of intervention
  Carotid-femoral pulse wave velocity (PWV), a preclinical marker of cardiovascular disease (CVD), is measured in meters per second (m/s) using applanation tonometry (SphygmoCor, AtCor Medical). Participants are positioned supine on a padded exam table after resting quietly for approximately five minutes. Brachial blood pressure is measured in millimeters of mercury (mmHg) using an automated cuff device. Pressure waveforms are recorded at the carotid artery (neck) and femoral artery (upper leg) using a handheld tonometer. The time delay between carotid and femoral pulse waves is used to calculate PWV, an indicator of arterial stiffness. The procedure is non-invasive and typically requires approximately five minutes to complete.
Glucose (mg/dL) | Baseline and after 4 weeks of intervention
  After a 10- to 12-hour overnight fast, participants undergo a 2-hour oral glucose tolerance test (OGTT) at the Clinical Research Unit, SUNY Upstate Medical University. Venous blood samples are collected at -15, 0, 30, 60, 90, and 120 minutes relative to glucose ingestion. At time 0 minutes, participants consume a commercially prepared standard 75-gram glucose solution; youth participants receive 1.75 grams of glucose per kilogram of body weight, not exceeding 75 grams total. After the final blood collection at 120 minutes, participants are provided a snack and continue their study visit. Blood is collected in pre-chilled aprotinin/EDTA tubes and processed for analysis of glucose (mg/dL).
Insulin (μIU/mL) | Baseline and after 4 weeks of intervention
  After a 10- to 12-hour overnight fast, participants undergo a 2-hour oral glucose tolerance test (OGTT) at the Clinical Research Unit, SUNY Upstate Medical University. Venous blood samples are collected at -15, 0, 30, 60, 90, and 120 minutes relative to glucose ingestion. At time 0 minutes, participants consume a commercially prepared standard 75-gram glucose solution; youth participants receive 1.75 grams of glucose per kilogram of body weight, not exceeding 75 grams total. After the final blood collection at 120 minutes, participants are provided a snack and continue their study visit. Blood is collected in pre-chilled aprotinin/EDTA tubes and processed for analysis of insulin (μIU/mL).
C-peptide (ng/mL) | Baseline and after 4 weeks of intervention
  After a 10- to 12-hour overnight fast, participants undergo a 2-hour oral glucose tolerance test (OGTT) at the Clinical Research Unit, SUNY Upstate Medical University. Venous blood samples are collected at -15, 0, 30, 60, 90, and 120 minutes relative to glucose ingestion. At time 0 minutes, participants consume a commercially prepared standard 75-gram glucose solution; youth participants receive 1.75 grams of glucose per kilogram of body weight, not exceeding 75 grams total. After the final blood collection at 120 minutes, participants are provided a snack and continue their study visit. Blood is collected in pre-chilled aprotinin/EDTA tubes and processed for analysis of C-peptide (ng/mL).
Total glucagon-like peptide-1 (GLP-1) (pmol/L) | Baseline and after 4 weeks of intervention
  After a 10- to 12-hour overnight fast, participants undergo a 2-hour oral glucose tolerance test (OGTT) at the Clinical Research Unit, SUNY Upstate Medical University. Venous blood samples are collected at -15, 0, 30, 60, 90, and 120 minutes relative to glucose ingestion. At time 0 minutes, participants consume a commercially prepared standard 75-gram glucose solution; youth participants receive 1.75 grams of glucose per kilogram of body weight, not exceeding 75 grams total. After the final blood collection at 120 minutes, participants are provided a snack and continue their study visit. Blood is collected in pre-chilled aprotinin/EDTA tubes and processed for analysis of total glucagon-like peptide-1 (GLP-1) (pmol/L).
Glucose-dependent insulinotropic polypeptide (GIP) (pg/mL) | Baseline and after 4 weeks of intervention
  After a 10- to 12-hour overnight fast, participants undergo a 2-hour oral glucose tolerance test (OGTT) at the Clinical Research Unit, SUNY Upstate Medical University. Venous blood samples are collected at -15, 0, 30, 60, 90, and 120 minutes relative to glucose ingestion. At time 0 minutes, participants consume a commercially prepared standard 75-gram glucose solution; youth participants receive 1.75 grams of glucose per kilogram of body weight, not exceeding 75 grams total. After the final blood collection at 120 minutes, participants are provided a snack and continue their study visit. Blood is collected in pre-chilled aprotinin/EDTA tubes and processed for analysis of glucose-dependent insulinotropic polypeptide (GIP) (pg/mL).
Leptin (ng/mL) | Baseline and after 4 weeks of intervention
  After a 10- to 12-hour overnight fast, participants undergo a 2-hour oral glucose tolerance test (OGTT) at the Clinical Research Unit, SUNY Upstate Medical University. Venous blood samples are collected at -15, 0, 30, 60, 90, and 120 minutes relative to glucose ingestion. At time 0 minutes, participants consume a commercially prepared standard 75-gram glucose solution; youth participants receive 1.75 grams of glucose per kilogram of body weight, not exceeding 75 grams total. After the final blood collection at 120 minutes, participants are provided a snack and continue their study visit. Blood is collected in pre-chilled aprotinin/EDTA tubes and processed for analysis of leptin (ng/mL).
Adiponectin (μg/mL) | Time Frame: Baseline and after 4 weeks of intervention
  After a 10- to 12-hour overnight fast, participants undergo a 2-hour oral glucose tolerance test (OGTT) at the Clinical Research Unit, SUNY Upstate Medical University. Venous blood samples are collected at -15, 0, 30, 60, 90, and 120 minutes relative to glucose ingestion. At time 0 minutes, participants consume a commercially prepared standard 75-gram glucose solution; youth participants receive 1.75 grams of glucose per kilogram of body weight, not exceeding 75 grams total. After the final blood collection at 120 minutes, participants are provided a snack and continue their study visit. Blood is collected in pre-chilled aprotinin/EDTA tubes and processed for analysis of adiponectin (μg/mL).
Ghrelin (pg/mL) | Baseline and after 4 weeks of intervention
  After a 10- to 12-hour overnight fast, participants undergo a 2-hour oral glucose tolerance test (OGTT) at the Clinical Research Unit, SUNY Upstate Medical University. Venous blood samples are collected at -15, 0, 30, 60, 90, and 120 minutes relative to glucose ingestion. At time 0 minutes, participants consume a commercially prepared standard 75-gram glucose solution; youth participants receive 1.75 grams of glucose per kilogram of body weight, not exceeding 75 grams total. After the final blood collection at 120 minutes, participants are provided a snack and continue their study visit. Blood is collected in pre-chilled aprotinin/EDTA tubes and processed for analysis of ghrelin (pg/mL).
C-reactive protein (CRP) (mg/L) | Baseline and after 4 weeks of intervention
  After a 10- to 12-hour overnight fast, participants undergo a 2-hour oral glucose tolerance test (OGTT) at the Clinical Research Unit, SUNY Upstate Medical University. Venous blood samples are collected at -15, 0, 30, 60, 90, and 120 minutes relative to glucose ingestion. At time 0 minutes, participants consume a commercially prepared standard 75-gram glucose solution; youth participants receive 1.75 grams of glucose per kilogram of body weight, not exceeding 75 grams total. After the final blood collection at 120 minutes, participants are provided a snack and continue their study visit. Blood is collected in pre-chilled aprotinin/EDTA tubes and processed for analysis of C-reactive protein (CRP) (mg/L).
Interleukin-6 (IL-6) (pg/mL) | Baseline and after 4 weeks of intervention
  After a 10- to 12-hour overnight fast, participants undergo a 2-hour oral glucose tolerance test (OGTT) at the Clinical Research Unit, SUNY Upstate Medical University. Venous blood samples are collected at -15, 0, 30, 60, 90, and 120 minutes relative to glucose ingestion. At time 0 minutes, participants consume a commercially prepared standard 75-gram glucose solution; youth participants receive 1.75 grams of glucose per kilogram of body weight, not exceeding 75 grams total. After the final blood collection at 120 minutes, participants are provided a snack and continue their study visit. Blood is collected in pre-chilled aprotinin/EDTA tubes and processed for analysis of

CONTACTS AND LOCATIONS:
Locations (1):
- Syracuse University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-10-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT07215533/Prot_000.pdf
  • Informed Consent Form (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT07215533/ICF_001.pdf